CLINICAL TRIAL: NCT06010979
Title: Clinical Cohort Study of Knee Arthroplasty Assisted by Digital Technology
Status: Recruiting | Type: Observational
Sponsor: Tian Hua (Other)
Responsible Party: Sponsor-Investigator, Tian Hua, archiater, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: TKAcohort
Record Dates: First submitted 2023-08-09; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; knee osteoarthritis; computer navigation; robotic system; patient-spercific instrumentation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- conventional group: Conventional instrument-assisted knee arthroplasty
  Interventions: Procedure: conventional intrumentation assisted knee arthroplasty
- CAS group: computer navigation assisted knee arthroplasty
  Interventions: Procedure: computer navigation assisted knee arthroplasty
- RAS group: robotic system assisted knee arthroplasty
  Interventions: Procedure: robotic system assisted knee arthroplasty
- PSI group: patient-spercific instrumentation assisted knee arthroplasty
  Interventions: Procedure: patient-spercific assisted knee arthroplasty

INTERVENTIONS:
Procedure: conventional intrumentation assisted knee arthroplasty — conventional intrumentation assisted knee arthroplasty
  Groups: conventional group
Procedure: computer navigation assisted knee arthroplasty — computer navigation assisted knee arthroplasty
  Groups: CAS group
Procedure: robotic system assisted knee arthroplasty — robotic system assisted knee arthroplasty
  Groups: RAS group
Procedure: patient-spercific assisted knee arthroplasty — patient-spercific assisted knee arthroplasty
  Groups: PSI group

SUMMARY:
Through this cohort study, previous clinical data can be systematically reviewed and supplemented through clinical follow-up. Prospective enrollment and follow-up observation of subsequent patients can also be carried out to build a retrospective-prospective two-way cohort study. The intraoperative, perioperative, clinical follow-up and health economics of surgical robot, computer navigation, personalized osteotomy guide and other digital technologies and traditional TKA were comprehensively and objectively compared, the results and conclusions of the center were summarized and reported, and the effectiveness and safety of digital assistive technology applied to TKA were explored, providing references for clinical diagnosis and follow-up research.

DETAILED DESCRIPTION:
Through this cohort study, previous clinical data can be systematically reviewed and supplemented by follow-up visits. Prospective enrollment and follow-up of subsequent patients can also be carried out to build a retrospective-prospective two-way cohort study. The preoperative situation (general statistical information, educational level, preoperative clinical function score, etc.), intraoperative situation (operative time, intraoperative blood loss, intraoperative complications, etc.), perioperative situation (total postoperative blood loss, blood transfusion rate, postoperative complications, etc.) and clinical follow-up situation were comprehensively and objectively compared with surgical robot, computer navigation, personalized osteotomy guide and other digital technologies and traditional TKA We summarized and reported the results and conclusions of the center (postoperative force line, implant location, pain, mobility, clinical function score, patient satisfaction and postoperative complications, etc.) and health economics (average length of stay, hospitalization cost, etc.) to provide reference for clinical diagnosis and follow-up research.

ELIGIBILITY:
Inclusion Criteria:

* a. primary knee osteoarthritis;
* b. Unilateral primary knee replacement;
* c. Surgical methods were traditional surgery, surgical robot, computer navigation or personalized osteotomy guide

Exclusion Criteria:

* a. A history of renal insufficiency (Cr > 2.5), liver insufficiency, severe heart disease (or coronary stenting within the last 12 months), severe respiratory disease, history of VTE or high risk of thrombosis (hereditary/acquired thrombotic disease), cotting disorder, stroke, and malignancy;
* b. Those who do not accept this test for any reason and refuse to sign the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing knee replacement in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mechanical axis | Postoperative day 3
  The postoperative HKA Angle was measured, that is, the Angle between the center of the hip joint and the center of the knee joint and the center of the knee joint and the center of the ankle joint on the full-length X-ray film of the lower limb. The target Angle was defined as 0°, the Angle was positive when the knee was varus, the Angle was negative when the knee was varus, and the acceptable range was ±3°, beyond which the line deviation was defined.

SECONDARY OUTCOMES:
operation time | immediately after the surgery
  The surgical time is defined as the time from incision to the completion of the skin suture, accurate to minutes
Intraoperative blood loss | immediately after the surgery
  Intraoperative blood loss = total amount of fluid drawn during the operation - intraoperative irrigation volume + intraoperative gauze infiltration blood loss, accurate to ml
Intraoperative complications | immediately after the surgery
  Various complications occurred during the operation were recorded
Total postoperative blood loss | Postoperative day 3
  Gross linear equation was used to calculate total blood loss and latent blood loss 3 days after surgery. Total blood loss = preoperative blood volume (PBV) × (preoperative hematocrit - postoperative hematocrit). PBV was calculated using Nadler method: PBV=K1× height (m) 3+K2× weight (kg) +K3, where male K1=0.3669, K2=0.03219, K3=0.6041; Female K1=0.3561, K2=0.03308, K3=0.1833. Postoperative total blood loss = total blood loss - intraoperative blood loss;
Blood transfusion rate | At discharge
  The postoperative blood transfusion situation and the amount of blood transfusion were recorded. The blood was transfused mainly with suspended red blood cells, and the amount of a single transfusion was 400ml. The Hb situation was evaluated again by blood routine review on the morning of the second day after transfusion.
  Indications for postoperative blood transfusion: No blood transfusion for Hb up to 8g/L or above; Hb up to 7g/L (including) must be transfused; Hb is between 7-8g/L, and blood transfusion should be given when anemia symptoms such as dizziness, weakness, palpitation, etc.
Postoperative complication | 3 years postoperatively
  The postoperative complications such as wound nonunion, wound infection, hematomas and anemia were recorded.
Rotation Angle of femur prosthesis | Postoperative day 3
  On the horizontal plane of CT scan of the affected knee, the Angle between the line of the posterior condyle of the femoral prosthesis and the line of the transcondyle of the femur was shown. The target Angle was defined as 0° external rotation of the femoral prosthesis, positive Angle during external rotation, negative Angle during internal rotation, acceptable range of ±2°, beyond which was defined as angular deviation
Visual analogue scale | Postoperative day 3
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 2 weeks postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 6 weeks postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 3 months postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 6 months postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 12 months postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 24 months postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Visual analogue scale | 36 months postoperatively
  The pain of the affected limb was assessed by Visual analogue scale. The highest score is ten and the lowest score is zero. A higher score indicates a higher level of pain.
Range of motion | 3 days postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 2 weeks postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 6 weeks postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 3 months postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 6 months postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 12 months postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 24 months postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
Range of motion | 36 months postoperatively
  The Range of motion of the knee on the operative side of the patient was measured
knee society score | 6 weeks postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
knee society score | 3 months postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
knee society score | 6 months postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
knee society score | 12 months postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
knee society score | 24 months postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
knee society score | 36 months postoperatively
  This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. The evaluation was numerically quantified (see table), and the knee joint score and the functional score were obtained respectively. The higher the value, the better the function.
Western Ontario and McMaster Universities Osteoarthritis Index | 6 weeks postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Western Ontario and McMaster Universities Osteoarthritis Index | 3 months postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Western Ontario and McMaster Universities Osteoarthritis Index | 6 months postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Western Ontario and McMaster Universities Osteoarthritis Index | 12 months postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Western Ontario and McMaster Universities Osteoarthritis Index | 24 months postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Western Ontario and McMaster Universities Osteoarthritis Index | 36 months postoperatively
  This score is used to assess the severity of arthritis and its therapeutic effect based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. A higher score indicates better functionality.
Patient satisfaction | 6 months postoperatively
  At follow-up, patients' satisfaction scores were recorded (using 5-Likert scale). The higher the score, the higher the satisfaction
Patient satisfaction | 12 months postoperatively
  At follow-up, patients' satisfaction scores were recorded (using 5-Likert scale). The higher the score, the higher the satisfaction
Patient satisfaction | 24 months postoperatively
  At follow-up, patients' satisfaction scores were recorded (using 5-Likert scale). The higher the score, the higher the satisfaction
Patient satisfaction | 36 months postoperatively
  At follow-up, patients' satisfaction scores were recorded (using 5-Likert scale). The higher the score, the higher the satisfaction
Length of stay | an average of 3 days postoperatively
  The number of days a patient stays in hospital from admission to discharge
Medical expenses | an average of 3 days postoperatively
  The total cost of a patient from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Tian Hua, MD, Study Director — Director
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
It will be published as an academic paper
Supporting Information: Study Protocol, CSR
Time Frame: When data collection is complete
Access Criteria: All the researchers who need it